CLINICAL TRIAL: NCT01848275
Title: The Clinical Efficacy Comparison of Two Renal Sympathetic Denervation Strategies ---- Full Length Versus Proximal Renal Arteries Ablation
Brief Title: Full Length Versus Proximal Renal Arteries Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN- RDN Strategy
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Group 1 received ablation from distal to ostial of bilateral renal arteries
  Interventions: Device: Thermocool®Rcatheter
- Group 2 (Experimental): group 2 received ablation at proximal of bilateral renal arteries
  Interventions: Device: Thermocool®Rcatheter

INTERVENTIONS:
Device: Thermocool®Rcatheter — The full length RDN was performed discretely from distal to proximal by point to point using Thermocool®Rcatheter
  Arms: Group 1
Device: Thermocool®Rcatheter — The proximity renal denervation was performed discretely at 10-15 mm of proximal renal artery, using Thermocool®Rcatheter
  Arms: Group 2

SUMMARY:
Catheter-based renal sympathetic modification has been documented to be effective option for blood pressure control in patients with resistant hypertension, but the safety is still concerned around worldwide. Based on anatomic findings, blocking renal sympathetic nerves at proximity may be enough for successful renal sympathetic modifications. This study was designed to compare the efficacy and safety of full length versus proximal ablation of bilateral renal arteries.

DETAILED DESCRIPTION:
After baseline assessment was completed, patients with resistant hypertension were enrolled, and randomly divided into two groups. This study is going to recruit 40 patients (group 1 VS group 2 = 1:1) with a follow-up duration of one year. Group 1 received ablation from distal to ostial of bilateral renal arteries, group 2 received ablation at proximal of bilateral renal arteries. RDN was performed with saline irrigated catheter. Office and ambulatory blood pressure was measured.

ELIGIBILITY:
Inclusion Criteria:

* office systolic blood pressure of 160 mm Hg or more,
* patients had to be on a stable drug regimen of at least 3 antihypertensive medications with no changes for 1 month before enrollment.
* Despite being treated with at least three antihypertensive drugs(including one diuretic), or confirmed intolerance to medications;
* ≥ 18 years old,;
* did not have any known secondary cause of hypertension;
* had a glomerular filtration rate estimated with the modification of diet in renal disease formula, of 45 ml/min/1.73m2 or more.

Exclusion Criteria:

* patients with type 1 diabetes,
* implanted pacemakers or implantable cardioverter defibrillators;
* pregnant women;
* haemodynamically significant valvular disease;
* patients with renovascular abnormalities(including mild to severe renal artery stenosis, especially caused by atherosclerosis, previous renal stenting or angioplasty, or known dual renal arteries, or diameter of renal artery identified by angiography less than 4 mm and/or length of renal artery less than 2 cm)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | one year
  office BP and Ambulatory blood pressure

SECONDARY OUTCOMES:
ablation-related complications | one year
  ablation-related complications such as pseudoaneurysm，renal artery injury

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China